CLINICAL TRIAL: NCT01662895
Title: Futility Study of Deferoxamine in Intracerebral Hemorrhage
Brief Title: High-Dose Deferoxamine in Intracerebral Hemorrhage
Acronym: HI-DEF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: By DSMB on October 18, 2013 due to increased incidence of ARDS. See modified protocol [NCT02175225
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Medical University of South Carolina (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Massachusetts General Hospital (Other); Tufts Medical Center (Other); University of Massachusetts, Worcester (Other); University of Pennsylvania (Other); Johns Hopkins University (Other); University of Maryland (Other); University of Virginia (Other); Duke University (Other); University of North Carolina (Other); University of Florida (Other); The Cleveland Clinic (Other); Henry Ford Hospital (Other); Ohio State University (Other); St. Joseph's Hospital and Medical Center, Phoenix (Other); University of California, San Francisco (Other); Oregon Health and Science University (Other); Yale New Haven Hospital (Unknown); University of Iowa (Other); Hartford Hospital (Other); The University of Texas Health Science Center, Houston (Other); Rhode Island Hospital (Other); Stanford University (Other); University of Washington (Other); University of Calgary (Other); Hopital de l'Enfant-Jesus (Other); University of Alberta (Other); Dalhousie University (Other)
Responsible Party: Principal Investigator, Magdy Selim, Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012P-000005; U01NS074425 (NIH)
Record Dates: First submitted 2012-07-30; First posted 2012-08-13 (Estimated); Results first posted 2019-05-30 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Intracerebral Hemorrhage
Keywords: Brain hemorrhage; Cerebral Hemorrhage; Deferoxamine; Hi-DEF Trial
MeSH Terms: conditions — Cerebral Hemorrhage; Intracranial Hemorrhages | interventions — Deferoxamine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deferoxamine (Active Comparator): Deferoxamine mesylate supplied in vials containing 2 gm of sterile, lyophilized, powdered deferoxamine mesylate. The drug will be reconstituted for injection, by dissolving in 20 ml of sterile water. The reconstituted drug will be further diluted in normal saline to achieve a final concentration of 7.5 mg per ml.
  Interventions: Drug: Deferoxamine
- Normal Saline (Placebo Comparator): 0.9% sodium chloride
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Deferoxamine — Deferoxamine mesylate(62 mg/kg/day up to a maximum daily dose of 6000 mg/day) given by a continuous IV infusion for 5 consecutive days beginning within 24 hours of ICH symptom onset.
  Other Names: Deferoxamine Mesylate
  Arms: Deferoxamine
Drug: Normal saline — This is a placebo. Normal saline will be given by a continuous IV infusion for 5 consecutive days beginning within 24 hours of ICH symptom onset.
  Other Names: 0.90% Sodium Chloride Solution
  Arms: Normal Saline

SUMMARY:
The main purpose of this study is to determine whether treatment with deferoxamine mesylate is of sufficient promise to improve outcome before pursuing a larger clinical trial to examine its effectiveness as a treatment for brain hemorrhage.

DETAILED DESCRIPTION:
Several studies show that hemoglobin breakdown and subsequent iron accumulation in the brain play a role in mediating secondary neuronal injury after intracerebral hemorrhage (ICH); and that treatment with the iron chelator, deferoxamine (DFO), provides neuroprotection in animal models of ICH. The investigators recently concluded a phase-I, safety and dose-finding study of DFO in patients with ICH; repeated daily intravenous (IV) infusions of DFO in doses up to 62 mg/kg/day (up to a maximum daily dose of 6000 mg/day) were well-tolerated and did not increase serious adverse events or mortality. The current study builds on these results to assess the potential utility of DFO as a therapeutic intervention in ICH.

This is a prospective, multi-center, double-blind, randomized, placebo-armed, phase-II, futility clinical study to determine if this maximum tolerated dose of DFO is of sufficient promise to improve outcome prior to embarking on a large-scale and costly phase III study to assess its efficacy in ICH. The investigators will randomize 324 subjects with ICH equally (1:1) to either DFO at 62 mg/kg/day (up to a maximum daily dose of 6000 mg/day), or saline placebo, given by continuous IV infusion for 5 consecutive days. Treatment will be initiated within 24 hours after ICH symptom onset. Subjects will be stratified based on baseline ICH score (0-2 vs. 3-5) and ICH onset-to-treatment time (OTT) window (≤12h vs. >12-24h), so that the resulting randomization ratio is 1:1 within each ICH score and OTT window strata.

The main objectives are:

1. To assess whether it would be futile to move DFO forward into a Phase III trial based on the end point of good outcome (defined as dichotomized modified Rankin Scale score of 0-2 at 3 months). At the conclusion of the study, the proportion of DFO-treated subjects with a good outcome will be compared to the placebo proportion in a futility analysis. If the DFO-treated proportion is less than 12% greater than the placebo proportion, then it would be futile to move DFO forward to future Phase III testing.
2. To collect more data on treatment-related adverse events in order to ascertain that patients with ICH can tolerate this dose given over an extended 5-day duration of infusion without experiencing unreasonable neurological complications, increased mortality, or other serious adverse events related to DFO use.

Secondary and exploratory objectives include:

1- Determining the overall distribution of scores on mRS at 3 months in DFO-treated subjects, and to perform a dichotomized analysis considering the proportion of DFO- and placebo-treated subjects with mRS 0-3.

Successful completion of this study will provide a crucial "go/no-go" signal for DFO in ICH. Futility will discourage a major phase III trial, whereas non-futility will offer strong support for a phase III study to detect clinical efficacy. Results from this study can provide valuable information to guide the design and sample size estimation of a potential future Phase III trial. ICH is a frequent cause of disability and death. A successful study demonstrating the efficacy of DFO would be of considerable public health significance.

Update: Enrollment into the trial was terminated by the Data and Safety Monitoring Board because of an imbalance in subjects with reported ARDS. At the time of termination, 42 subjects had been enrolled. As a result, any formal evaluation of these objectives would be under-powered, but descriptive statistics are provided. The protocol was subsequently modified to protect subject safety, and the trial was re-initiated as iDEF (NCT02175225).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 80 years
2. The diagnosis of ICH is confirmed by brain CT scan
3. NIHSS score ≥ 6 and GCS > 6 upon presentation
4. The first dose of the study drug can be administered within 24h of ICH symptom onset
5. Functional independence prior to ICH, defined as pre-ICH mRS ≤ 1
6. Signed and dated informed consent is obtained.

Exclusion Criteria:

1. Previous chelation therapy or known hypersensitivity to DFO products
2. Known severe iron deficiency anemia (defined as hemoglobin concentration < 7g/dL or requiring blood transfusions)
3. Abnormal renal function, defined as serum creatinine > 2 mg/dL
4. Planned surgical evacuation of ICH prior to administration of study drug (placement of a catheter for ventricular drainage is not a contraindication to enrollment)
5. Suspected secondary ICH related to tumour, ruptured aneurysm or arteriovenous malformation, hemorrhagic transformation of an ischemic infarct, or venous sinus thrombosis
6. Infratentorial hemorrhage
7. Irreversibly impaired brainstem function (bilateral fixed and dilated pupils and extensor motor posturing)
8. Complete unconsciousness, defined as a score of 3 on item 1a of the NIHSS (Responds only with reflex motor or autonomic effects or totally unresponsive, and flaccid)
9. Pre-existing disability, defined as pre-ICH mRS ≥ 2
10. Coagulopathy - defined as elevated aPTT or INR >1.3 upon presentation; concurrent use of direct thrombin inhibitors (such as dabigatran), direct factor Xa inhibitors (such as rivaroxaban), or low-molecular-weight heparin
11. Taking iron supplements containing ≥ 325 mg of ferrous iron, or prochlorperazine
12. Patients with heart failure taking > 500 mg of vitamin C daily
13. Known severe hearing loss
14. Known pregnancy, or positive pregnancy test, or breastfeeding
15. Patients known or suspected of not being able to comply with the study protocol due to alcoholism, drug dependency, noncompliance, living in another state or any other cause
16. Positive drug screen for cocaine upon presentation
17. Any condition which, in the judgement of the investigator, might increase the risk to the patient
18. Life expectancy of less than 90 days due to comorbid conditions
19. Concurrent participation in another research protocol for investigation of another experimental therapy
20. Indication that a new Do Not Resuscitate (DNR) or Comfort Measures Only (CMO) order will be implemented within the first 72 hours of hospitalization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-03-18 (Actual); Primary Completion 2014-01-15 (Actual); Study Completion 2018-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Magdy Selim, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center/Harvard Medical School
Locations (29):
- United States (25):
  - St. Joseph's Hospital, Phoenix, Arizona
  - Stanford University Hospital, Palo Alto, California
  - San Francisco General Hospital, San Francisco, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - The University of Florida College of Medicine, Jacksonville, Florida
  - University of Iowa Hospital, Iowa City, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - The University of Texas Health Science Center, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Harborview Medical Center, Seattle, Washington
- Canada (4):
  - Foothills Medical Center, Calgary, Alberta
  - Mackenzie Health Sciences Centre, Edmonton, Alberta
  - Halifax Infirmary, Halifax, Nova Scotia
  - Hôpital de l'Enfant-Jésus - CHU de Québec, Québec

REFERENCES:
- [Background] Selim M. Deferoxamine mesylate: a new hope for intracerebral hemorrhage: from bench to clinical trials. Stroke. 2009 Mar;40(3 Suppl):S90-1. doi: 10.1161/STROKEAHA.108.533125. Epub 2008 Dec 8. PMID 19064798
- [Background] Selim M, Yeatts S, Goldstein JN, Gomes J, Greenberg S, Morgenstern LB, Schlaug G, Torbey M, Waldman B, Xi G, Palesch Y; Deferoxamine Mesylate in Intracerebral Hemorrhage Investigators. Safety and tolerability of deferoxamine mesylate in patients with acute intracerebral hemorrhage. Stroke. 2011 Nov;42(11):3067-74. doi: 10.1161/STROKEAHA.111.617589. Epub 2011 Aug 25. PMID 21868742
- [Background] Gu Y, Hua Y, Keep RF, Morgenstern LB, Xi G. Deferoxamine reduces intracerebral hematoma-induced iron accumulation and neuronal death in piglets. Stroke. 2009 Jun;40(6):2241-3. doi: 10.1161/STROKEAHA.108.539536. Epub 2009 Apr 16. PMID 19372448
- [Background] Okauchi M, Hua Y, Keep RF, Morgenstern LB, Xi G. Effects of deferoxamine on intracerebral hemorrhage-induced brain injury in aged rats. Stroke. 2009 May;40(5):1858-63. doi: 10.1161/STROKEAHA.108.535765. Epub 2009 Mar 12. PMID 19286595
- [Derived] Roh DJ, Poyraz FC, Mao E, Shen Q, Kansara V, Cottarelli A, Song S, Nemkov T, Kumar A, Hudson KE, Ghoshal S, Park S, Agarwal S, Connolly ES, Claassen J, Kreuziger LB, Hod E, Yeatts S, Foster LD, Selim M. Anemia From Inflammation After Intracerebral Hemorrhage and Relationships With Outcome. J Am Heart Assoc. 2024 Jul 16;13(14):e035524. doi: 10.1161/JAHA.124.035524. Epub 2024 Jul 9. PMID 38979830
- [Derived] Yeatts SD, Palesch YY, Moy CS, Selim M. High dose deferoxamine in intracerebral hemorrhage (HI-DEF) trial: rationale, design, and methods. Neurocrit Care. 2013 Oct;19(2):257-66. doi: 10.1007/s12028-013-9861-y. PMID 23943316

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Deferoxamine | Normal Saline
Started | 21 | 21
Initiated Study Drug | 21 | 21
Completed | 21 | 20
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deferoxamine | Normal Saline | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Median (Full Range); unit: years] | 64 [35 to 77] | 64 [43 to 77] | 64 [35 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 14 | 12 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 20 | 19 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 15 | 17 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Modified Rankin Scale (mRS) Score 0-2
Description: The primary outcome measure of efficacy is the modified Rankin Scale (mRS) score, dichotomized to define good functional outcome as mRS 0-2 at 90 days.
  The minimum mRS score is 0 (i.e. no disability). The maximum score is 6 (i.e. dead).
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine | Normal Saline
Number analyzed (Participants) | 21 | 20
Participants | 6 | 10

2. Secondary Outcome: Number of Subjects With mRS Score 0-3
Description: The proportion of DFO- and placebo-treated subjects with mRS 0-3 vs. 4-6 at 90 days
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine | Normal Saline
Number analyzed (Participants) | 21 | 20
Participants | 12 | 14

3. Other Pre Specified Outcome: Number of Subjects With Allergic/Anaphylactic Reaction
Time Frame: within 7 days or discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine | Normal Saline
Number analyzed (Participants) | 21 | 21
Participants | 0 | 0

4. Other Pre Specified Outcome: Number of Patients With Hypotension
Time Frame: within 7 days or discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine | Normal Saline
Number analyzed (Participants) | 21 | 21
Participants | 1 | 1

5. Other Pre Specified Outcome: Number of Patients With New Visual or Auditory Changes
Time Frame: within 7 days or discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine | Normal Saline
Number analyzed (Participants) | 21 | 21
Participants | 0 | 1

6. Other Pre Specified Outcome: Number of Patients With Serious Adverse Events
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine | Normal Saline
Number analyzed (Participants) | 21 | 21
Participants | 9 | 6

7. Other Pre Specified Outcome: Number of Patients Who Died During the 90-day Study Period
Description: Mortality at any time from randomization through day-90
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine | Normal Saline
Number analyzed (Participants) | 21 | 21
Participants | 3 | 0

8. Post Hoc Outcome: Number of Subjects With Acute Respiratory Distress Syndrome
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine | Normal Saline
Number analyzed (Participants) | 21 | 21
Participants | 6 | 0

ADVERSE EVENTS:
Time Frame: All adverse events (serious and non-serious) were assessed until day-7 or discharge, whichever occurs earlier, and serious adverse events until day-90 (i.e. completion of the study) or withdrawal of consent.
Arm/Group | Deferoxamine | Normal Saline
All-Cause Mortality (participants affected / at risk) | 3/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 9/21 | 6/21
Other Adverse Events (participants affected / at risk) | 17/21 | 18/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferoxamine (N=21) | Normal Saline (N=21)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intracranial hypotension (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Neurological decompensation (Nervous system disorders) | 2 (3) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferoxamine (N=21) | Normal Saline (N=21)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Colour blindness acquired (Eye disorders) | 0 (0) | 1 (1)
Pupils unequal (Eye disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Infusion site erythema (General disorders) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Infusion site inflammation (General disorders) | 1 (1) | 0 (0)
Infusion site oedema (General disorders) | 1 (1) | 0 (0)
Infusion site pain (General disorders) | 1 (2) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 7 (7) | 6 (7)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4) | 4 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine abnormal (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Blood iron decreased (Investigations) | 2 (2) | 0 (0)
Blood magnesium increased (Investigations) | 1 (1) | 0 (0)
Blood urea abnormal (Investigations) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 1 (1)
Cardiac enzymes increased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Iron binding capacity total decreased (Investigations) | 1 (1) | 0 (0)
Prothrombin time (Investigations) | 1 (1) | 0 (0)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0)
Renal function test abnormal (Investigations) | 2 (2) | 0 (0)
Serum ferritin abnormal (Investigations) | 1 (1) | 0 (0)
Transferrin decreased (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Urine analysis abnormal (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Neurological decompensation (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 0 (0)
Ureteric dilatation (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Phlebitis (Vascular disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely, and only 42 subjects were enrolled. As a result, any formal evaluation of these outcomes would be under-powered. Only descriptive statistics are provided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No